CLINICAL TRIAL: NCT03117101
Title: An Open-label, Dose-finding Phase I Study to Determine the Maximum Tolerated Dose, Recommended Dose, Pharmacokinetics, Pharmacodynamics of the Dual -VEGFR-FGFR Tyrosine Kinase Inhibitor, AL3810, Givenorally as Single Agent to Patients With Advanced Solid Tumours
Brief Title: Study of the AL3810 in the Treatment of Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-80881-005
Record Dates: First submitted 2016-12-16; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Advanced Solid Tumors
Keywords: Tolerability Pharmacokinetics
MeSH Terms: interventions — E-3810; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation/ Dose extension of Lucitanib (Experimental): Dose escalation: Dose Level -1: 5 mg.Dose Level 1:.10 mg.Dose Level 2: 15 mg.Dose Level 3: 20 mg.
  Dose extension: Once the MTD was reached, the MTD-5 mg dose level was to be extended in order to enrol up to 12 patients (number of patients was to be determined regarding safety data) to better assess the toxicity profile, PK profile and antitumor activity.
  Interventions: Drug: Lucitanib

INTERVENTIONS:
Drug: Lucitanib
  Other Names: AL3810

SUMMARY:
This was a monocentric, open label, non-randomised, non-comparative, dose-finding phase I study

DETAILED DESCRIPTION:
Methodology:

This was a monocentric, open label, non-randomised, non-comparative, dose-finding phase I study with a traditional 3+3 design, conducted in Chinese patients with advanced solid tumours without an established therapeutic alternative.This study was performed in strict accordance with Good Clinical Practice including the archiving of essential documents.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female patient aged ≥ 18 years old and ≤ 70 years old.
2. Estimated life expectancy ≥ 12 weeks.
3. Histologically or cytologically confirmed, locally advanced or metastatic solid tumor, refractory to standard therapy or no standard therapy available.
4. Full recovery (to grade ≤ 1) from any prior surgical procedure(s) and from reversible side effects of prior therapy for cancer including radiation therapy, chemotherapy, small molecule therapeutics and immunotherapy.
5. Patients should be evaluable according to RECIST criteria, version 1.1.
6. Adequate haematological, hepatic and renal functions:

   Absolute neutrophil count (ANC) ≥ 1.5x 10^9/L Platelet counts ≥ 100 x 10^9/L. Haemoglobin ≥ 9 g/dL. Creatinine clearance > 50 mL/min (assessed with MDRD formula). Proteinuria qualitative test < 1+. If proteinuria qualitative test ≥ 1+, proteinuria over 24 hours should be < 1.0 g/24hrs.

   INR ≤ 1.5. AST, ALT ≤ 1.5 x Upper Limit of Normal Value (ULN) (≤ 3 x ULN in case of liver metastasis).

   Bilirubin < 1.5 x ULN.
7. Eastern Co-operative Group (ECOG) performance status ≤ 1.
8. Ability to swallow oral capsules.
9. Negative serum pregnancy test at screening in women of childbearing potential within 7 days prior the study drug intake.
10. Willingness and ability to comply with study procedures.
11. Signed written Informed Consent Form.

    Exclusion Criteria:
12. Participation in another therapeutic clinical trial at the same time or within 4 weeks prior to first AL3810 intake. In case of involvement in a non-interventional clinical trial (e.g. epidemiological study), inclusion in the present study is possible.
13. Foreseeable poor compliance to the study procedures.
14. Known active central nervous system (CNS) metastases not controlled by prior surgery or radiotherapy and/or low dose steroids.
15. Active second malignancy or history of other malignancy within 2 years, with the exception of non-melanoma skin cancers or carcinoma in situ (CIS) of the breast or cervix or controlled, superficial carcinoma of the bladder.
16. Chemotherapy including biologic/targeted therapy or immunological agents within 4 weeks or 5 half-lives of the agent, whichever the longest, before inclusion.
17. Previous treatment with bevacizumab within 3 months before the first day of AL3810 administration.
18. Patients who received radiotherapy within 4 weeks of starting study treatment.
19. Major surgery within 4 weeks before first day of study drug administration.
20. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification ≥ 3), angina, myocardial infarction or ventricular arrhythmia.
21. Significant cardiovascular disease or condition, including:

    Congestive heart failure requiring therapy. Ventricular and/or supra-ventricular arrhythmia requiring therapy. Severe conduction disturbance (including QTc interval prolongation > 450 msec [corrected], history of severe arrhythmia, or history of familial arrhythmia [e.g., Wolff-Parkinson-White syndrome]).

    Angina pectoris requiring therapy. Left ventricular ejection fraction (LVEF) < 50% evaluated by cardiac ultrasound (ECHO) or Multi Gated Acquisition Scan (MUGA).

    Myocardial infarction (MI) within 6 months prior to administration of the first dose.

    Cardiovascular disease > Class I, according to the New York Heart Association's (NYHA) Functional Criteria.

    Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg with optimized antihypertensive therapy or patients treated with ≥2 antihypertensive agents) or systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg with or without antihypertensive therapy.
22. Patients with thromboembolic events < 12 months prior to treatment start or at high risk of such events.
23. Ongoing treatment with warfarin or other oral anticoagulant.
24. Unavoidable concomitant treatment with any drug known for potential risk of causing Torsades de Pointes.
25. Serum potassium (K+) levels below LLN or 3.0 mmol/L at screening.
26. Patients who received administration of strong inhibitors of CYP2C8 and/or CYP3A4 or strong inducers of CYP3A4 within 7 days before the first dose of AL3810 or have on-going requirements for these medications (appendix 15).
27. Significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhoea associated with intestinal malabsorption, Crohn's disease, or decided by investigator.
28. Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, thyroid and adrenal gland.
29. Serious/active bacterial, viral or fungal infection (including known active human immunodeficiency virus [HIV] infection) requiring systemic treatment.
30. Concomitant uncontrolled severe systemic disease (e.g., uncontrolled diabetes mellitus, etc.).
31. Psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study procedures.
32. Known organ dysfunction which would either compromise the patient's safety or interfere with the evaluation of AL3810.
33. Men and women of child bearing potential unable or unwilling to employ effective contraception (abstinence, barrier method with spermicide, intrauterine device, or steroidal contraceptive for women and barrier method) during the study and for 6 months thereafter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Identify Dose-limiting toxicity (DLT) | 35 days
  To assess the tolerability of AL3810 in patients with advanced solid tumors
Identify maximum tolerated dose (MTD) | 35 days
  To assess the tolerability of AL3810 in patients with advanced solid tumors

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration) | Day0,Day8,Day15,Day22,Day29,Day57
  Metabolism profiling of AL3810 and its potential metabolites in plasma The potential food interaction on metabolism profile of AL 3810 in plasma
Tmax (time to maximum plasma concentration) | Day0,Day8,Day15,Day22,Day29,Day57
  Metabolism profiling of AL3810 and its potential metabolites in plasma The potential food interaction on metabolism profile of AL 3810 in plasma
AUC (area under the plasma concentration-time curve) | Day0,Day8,Day15,Day22,Day29,Day57
  Metabolism profiling of AL3810 and its potential metabolites in plasma The potential food interaction on metabolism profile of AL 3810 in plasma
Objective response rate (ORR) | 8 weeks
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion
progression free survival (PFS) | 8 weeks
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion
10.CBR (clinical benefit rate) | 8 weeks
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Fudan University; Junning Cao, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided